### **DOAC-CVT**

## Direct Oral Anticoagulants for the treatment of Cerebral Venous Thrombosis

#### Authors:

Mayte Sánchez van Kammen<sup>1</sup>, Anita van de Munckhof<sup>1</sup>, Jose M. Ferro<sup>2</sup>, Turgut Tatlisumak<sup>3</sup>, Jukka Putaala<sup>4</sup>, Jonathan M. Coutinho<sup>1</sup>

- 1. Department of Neurology, Amsterdam UMC, University of Amsterdam, Amsterdam, The Netherlands
- 2. Hospital da Luz, University of Lisbon, Lisbon, Portugal
- 3. Department of Clinical Neuroscience, Institute of Neuroscience and Physiology, Sahlgrenska Academy at University of Gothenburg and Department of Neurology, Sahlgrenska University Hospital, Gothenburg, Sweden
- 4. Department of Neurology, Helsinki University Hospital and University of Helsinki, Helsinki, Finland

# DIRECT ORAL ANTICOAGULANTS FOR THE TREATMENT OF CEREBRAL VENOUS THROMBOSIS: AN INTERNATIONAL PHASE IV STUDY

| Short title | DOAC-CVT |
|---------------------------|-----------------------------------|
| Version | 3.1 |
| Date | Update: 13-08-2024 |
| Project leader | Dr. Jonathan Coutinho |
| | Amsterdam UMC |
| | Email: j.coutinho@amsterdamumc.nl |
| Principal investigator(s) | See Appendix D |
| Sponsor | Amsterdam UMC |
| | Meibergdreef 9 |
| | 1105 AZ Amsterdam |
| Subsidising party | Trombosestichting Nederland |
| | Dobbeweg 1a |
| | 2254 AG Voorschoten |

#### **PROTOCOL SIGNATURE SHEET**

| Name | Signature | Date |
|-------------------------|-----------|------|
| Head of Department: | | |
| Prof.dr. D. van de Beek | | |
| Principal Investigator: | | |
| Dr. J. Coutinho | | |

#### **TABLE OF CONTENTS**

| 1. | INT | TRODUCTION AND RATIONALE | | |
|---|---|---|---|---|
| 2. | OB | ECTIVES | | 9 |
| 3. | STU | DY DESIGN | | 10 |
| 4. | STU | DY POPULATION | | 12 |
| | 4.1 | Population | | 12 |
| | 4.2 | Inclusion criteria | | 12 |
| | 4.3 | Exclusion criteria | | 12 |
| | 4.4 | Sample size calcu | lation | 12 |
| 5. | ME | HODS | | 14 |
| ; | 5.1 | Study parameters/ | /endpoints | 14 |
| | 5.1. | Primary study | endpoint | 14 |
| | 5.1. | Secondary stu | udy endpoints | 14 |
| ; | 5.2 | Study procedures. | | 15 |
| ; | 5.3 | Withdrawal of indiv | vidual subjects | 15 |
| ; | 5.4 | Premature termina | ation of the study | 15 |
| 6. | STA | TISTICAL ANALYS | SES | 16 |
| ( | 3.1 | Primary study end | point | 16 |
| | 6.1. | Main analysis | of primary endpoint | 16 |
| | 6.1. | Sensitivity and | alyses for the primary endpoint | 17 |
| | 6.1. | • . | alysis of primary endpoint | |
| ( | 3.2 | Secondary study p | parameter(s) | 18 |
| 7. | ETH | ICAL CONSIDERA | ATIONS | 19 |
| | 7.1 | Regulation statem | ent | 19 |
| | 7.2 | Recruitment and c | consent | 19 |
| | 7.3 | Benefits and risks | assessment | 19 |
| 8. | ADN | INISTRATIVE AS | PECTS, MONITORING AND PUBLICATION | 20 |
| | 3.1 | Handling and stora | age of data and documents | 20 |
| | 3.2 | Study Oversight | | 20 |
| | 3.3 | Public disclosure a | and publication policy | 22 |

#### **LIST OF ABBREVIATIONS**

CVT Cerebral venous thrombosis

VKA Vitamin K antagonists

DOAC Direct oral anticoagulants

VTE Venous thromboembolism

NIHSS National Institutes of Health Stroke Scale

MRV Magnetic resonance venography

ICH Intracranial hemorrhage

CNS Central nervous system

mRS Modified Rankin Scale

ISTH International Society on Thrombosis and Haemostasis

IRB Institutional Review Board

GDPR General Data Protection Regulation

eGFR Estimated glomerular filtration rate

Version 3.1 - 13-08-2024 5 of 31

#### **SUMMARY**

Rationale: Patients with cerebral venous thrombosis (CVT) are currently treated with anticoagulants during 3-12 months after diagnosis, to prevent worsening of the CVT and recurrent thrombosis, and to promote venous recanalization. Until recently, patients were generally treated with vitamin K antagonists (VKA). Direct oral anticoagulants (DOACs) are more practical in use than VKA and carry a lower risk of intracranial hemorrhage (ICH) in other conditions. One of the burning clinical questions is whether CVT patients can be safely treated with DOACs instead of VKA. In 2019, the first randomized trial on the safety and efficacy of DOACs in CVT was published (RESPECT-CVT). This exploratory study included 120 patients and the results suggest that DOACs can be safely used to treat CVT. Following RESPECT-CVT, use of DOACs to treat CVT is expected to rise, but given the limited sample size and strict selection criteria of RESPECT-CVT, additional data regarding the efficacy and safety of DOACs in CVT are required, especially from routine clinical care.

**Objective**: To assess the safety and efficacy of DOACs for the treatment of CVT in a real-world setting.

**Study design:** DOAC-CVT will be an international, prospective, comparative cohort study. We aim to recruit 1300 patients and anticipating a 3:2 ratio in DOAC:VKA use, we expect that in total 780 patients treated with a DOAC will be included.

**Study population:** Patients are eligible if they are >18 years old, have a radiologically confirmed CVT, and have started oral anticoagulant treatment (DOAC or VKA) within 30 days of CVT diagnosis.

**Primary study endpoint:** The primary endpoint is a composite of major bleeding (according to the criteria of the International Society on Thrombosis and Haemostasis) AND symptomatic recurrent venous thrombosis after 6 months of follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This is an observational study which poses no risk or burden to the participant. Only data that are collected as part of routine clinical care will be used.

ClinicalTrials.gov Identifier: NCT04660747

Version 3.1 - 13-08-2024 6 of 31

#### 1. INTRODUCTION AND RATIONALE

Cerebral venous thrombosis (CVT) is an uncommon thrombotic disorder that mainly affects young adults and children (Figure 1).<sup>1</sup> CVT often leads to severe neurological deficits, epileptic seizures, and decreased consciousness, and has a mortality rate of 5-15%.<sup>2,3</sup> A unique aspect of CVT is that the increased cerebral venous pressure leads to an intracerebral hemorrhage (ICH) in about 40% of patients.<sup>2</sup> Despite this high risk of major bleeding, anticoagulation is widely considered the main treatment for CVT, based on evidence from two small randomized trials.<sup>4</sup> Current guidelines recommend initial treatment with (low-molecular weight) heparin for 1-2 weeks, followed by vitamin K antagonists (VKA) for 3-12 months.<sup>5,6</sup>

Figure 1. T1-weighted MRI (A) and MR-venography (B) of a patient with superior sagittal sinus thrombosis.



A: Mid-sagittal T1 weighted MRI showing hyperintensity in the superior sagittal sinus, indicating fresh thrombus within the venous sinus (white arrows).

B: Sagittal MR-venogram of the same patient. There is absence of flow within the superior sagittal sinus, confirming there is a thrombosis in this vein (white arrows). There is normal opacification of the lateral sinus (black arrow).

One of the current burning clinical questions is whether CVT patients can be safely and effectively treated with direct oral anticoagulants (DOACs) instead of VKA. Apart from the practical advantages (stable dosing, no monitoring required), the substantially lower risk of ICH with DOACs compared to VKA in both venous thromboembolism and atrial fibrillation has sparked worldwide interest among neurologists.<sup>7,8</sup>

In 2019, the results of the first randomized trial on DOACs in CVT (RESPECT-CVT) were published.<sup>9</sup> The study was not powered for either superiority or non-inferiority, since it was clear from the start that such a large sample size would not be achievable in a disease as

Version 3.1 - 13-08-2024 7 of 31

rare as CVT. Nevertheless, the data of RESPECT-CVT indicate that dabigatran has a similar efficacy and safety as INR-adjusted warfarin for the treatment of CVT. A few small<sup>10,11</sup> and non-peer-reviewed<sup>12</sup> cohort studies have been published indicating results in the same direction.<sup>13</sup> Following the results of RESPECT-CVT, as well as the recent randomized SECRET-CVT trial and the retrospective ACTION-CVT study,<sup>14,15</sup> the use of DOACs to treat CVT is expected to rise. However, given the limited sample size and the strict inclusion and exclusion criteria of the randomized trials, additional data regarding the safety and efficacy of DOACs in CVT are much needed, especially data from routine clinical care.

DOAC-CVT will also provide more data on outcomes after CVT. While the mortality of CVT has decreased over the years,<sup>3</sup> several small-scale studies indicate that many CVT survivors suffer from chronic and debilitating symptoms, such as headache, fatigue, and concentration deficits.<sup>16,17</sup> The frequency and consistency of chronic symptoms in these studies suggest the existence of a "post-CVT syndrome", similar to the post-thrombotic syndrome seen in patients after a leg-vein thrombosis. While these studies clearly suggest that post-CVT syndrome commonly occurs, their small size limits the validity and generalizability of the data. The overall thrombotic recurrence rate after CVT is estimated at 5-10%,<sup>2,18</sup> which is lower than observed in other types of venous thromboembolism (VTE), but sufficiently powered, prospective, international studies are lacking. It is also unknown what the recurrence rate is according to the underlying risk profile, i.e. transient risk factors, persistent risk factors, and unprovoked thrombosis. More data about the post-CVT syndrome and long-term recurrence rate of VTE are urgently required, both for patient education and to guide future studies on how to mitigate this problem.

The main aim of the DOAC-CVT study (Direct oral anticoagulants for the treatment of cerebral venous thrombosis: an international phase IV study) will be to validate the efficacy and safety data of RESPECT-CVT in a real-world setting. Secondary aims are to investigate the frequency and burden of chronic post-CVT symptoms and the long-term thrombotic recurrence rate after CVT.

Version 3.1 - 13-08-2024 8 of 31

#### 2. OBJECTIVES

#### **Primary Objective**

To assess the safety and efficacy of DOACs vs. VKAs in patients with CVT, in terms of the 6-month risk of symptomatic recurrent VTE or major bleeding.

#### **Secondary Objectives**

In patients with CVT treated with DOACs vs. VKAs, to assess the 3, 6- and 12-month\*:

- All-cause mortality
- Symptomatic recurrent VTE rate
- Major bleeding rate
- Clinically relevant non-major bleeding rate
- Arterial thrombotic event rate
- Modified Rankin Scale score
- Oral anticoagulant cross-over rate with reasons for cross-over
- Cerebral venous recanalization rate at 6 months\*\*
- Frequency of chronic post-CVT symptoms at 12 months
- Thrombotic recurrence rate at 24 months
- \* 12-month follow-up: if performed as part of routine care
- \*\* Only in centers that perform 6-month follow-up imaging as part of routine clinical care

Version 3.1 - 13-08-2024 9 of 31

#### 3. STUDY DESIGN

DOAC-CVT is an international, prospective, phase IV, comparative observational cohort study. The study will use data that are collected as part of routine clinical care. It will be carried out during the course of 5 years in more than 60 hospitals worldwide with expertise in the treatment of CVT. Since this is an observational study, the choice of anticoagulant type and duration of treatment are left at the discretion of the treating physicians and patients. No treatment, intervention, or examinations are imposed on patients in the context of this study.

A blinded adjudication committee will evaluate the occurrence of the following endpoints: symptomatic recurrent VTE, major bleeding, clinically relevant non-major bleeding, arterial thrombotic events, and death (classified as cardiovascular, non-cardiovascular, or undetermined cause). Adjudication will be based on a standardized report form describing relevant clinical information and diagnostic test results, including slices of relevant imaging and local imaging reports. Using the available data, the adjudication committee will decide whether the registered event can be classified as a primary outcome (thrombotic or bleeding event). The adjudication committee will be blinded to the type of anticoagulant given (DOAC vs VKA).

Version 3.1 - 13-08-2024 10 of 31

Figure 2. Flowchart of baseline and follow-up time points and routine assessments at each time point\*



<sup>\*</sup>If part of routine care. Follow-up visits may be by phone or video

Version 3.1 - 13-08-2024 11 of 31

#### 4. STUDY POPULATION

#### 4.1 Population

Consecutive patients with CVT treated at the participating centres. Both patients who are admitted to the hospital and patients who are treated via outpatient clinic are eligible. A recruitment log will be kept by participating centers, which will also list non-included CVT patients with reasons of exclusion.

#### 4.2 Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

- Written informed consent for the use of observational data
- Age >18 years at the time of CVT diagnosis
- Radiologically confirmed CVT diagnosis (CT-venography, MRI or catheter angiography)
- Oral anticoagulant treatment (DOAC or VKA) started within 30 days of CVT diagnosis (patient may initially be treated with heparin)
- Inclusion in the study within 90 days of CVT diagnosis

#### 4.3 Exclusion criteria

As this is a phase IV study, the patient population should reflect routine clinical practice as much as possible. As such, the only exclusion criteria will be prevalent users and absolute contra-indications for the use of DOACs, i.e.:

- Anticoagulant treatment at the time of CVT diagnosis
- Pregnancy or lactation (post-partum women are eligible if they do not give breastfeeding)
- Mechanical heart valve
- Severe renal insufficiency (defined as an eGFR <15 ml/min)
- Severe liver disease resulting in clinically relevant coagulopathy

#### 4.4 Sample size calculation

DOAC-CVT is designed as a pragmatic exploratory phase IV study. Initially, DOAC-CVT was designed to recruit 500 patients in a three-year study period (until 15 January 2024). This convenience sample size was chosen because recruiting more patients was considered unfeasible due to the rarity of the disease. Now that international collaboration

Version 3.1 - 13-08-2024 12 of 31

and recruitment speed has exceeded expectations, recruitment in the DOAC-CVT study will continue for two additional years (until January 2026). As of January 2024, 635 patients have been recruited in the DOAC-CVT study. With an inclusion rate of approximately 30 patients per month, we expect to be able to recruit 1300 patients with CVT by the end of the study period in January 2026.

Version 3.1 - 13-08-2024 13 of 31

#### 5. METHODS

#### 5.1 Study parameters/endpoints

#### 5.1.1 Primary study endpoint

The primary endpoint is the composite of symptomatic recurrent VTE (i.e. recurrent CVT, DVT of any limb, pulmonary embolism, splanchnic vein, jugular, caval, renal, or catheter-related thrombosis) AND major bleeding (according to the criteria of the International Society on Thrombosis and Haemostasis [ISTH]<sup>19</sup>; see Appendix B) after 6 months of follow-up.

#### 5.1.2 Secondary study endpoints

Assessed at 3, 6 and 12 months\*:

- All-cause mortality
- Symptomatic recurrent VTE rate
- Major bleeding rate<sup>19</sup> (see Appendix B)
- Clinically relevant non-major bleeding rate<sup>20</sup> (see Appendix B)
- Arterial thrombotic event rate
- Modified Rankin Scale score
- Oral anticoagulant crossover rate with reasons for crossover

#### Assessed at 6 months\*\*:

 Cerebral venous recanalization rate – only if assessed as part of routine care

#### Assessed at 12 months\*:

- Frequency of chronic post-CVT symptoms

#### Assessed at 24 months:

- Symptomatic recurrent VTE rate

\* ± 1 month; 12-month follow-up only if performed as part of routine care

\*\* ± 2 months; cerebral venous recanalization will be scored according to the previously published Aguiar de Sousa classification<sup>21</sup> (see Appendix A)

Version 3.1 - 13-08-2024 14 of 31

#### 5.2 Study procedures

Baseline clinical and radiological data, treatment details, and events during primary admission will be collected for all patients. Participants will be followed-up at 3, 6, 12, and 24 months after diagnosis. This study will only analyse data that are collected as part of routine clinical care. Data collected during the 3-, 6-, and 12month follow-up visit include anticoagulant treatment details, imaging, clinical events, and functional outcome. Since not all hospitals perform a head MR with MRvenography or CT-venography at the 6-month follow-up visit as part of routine care, data on venous recanalization will be missing for some participating centers. Quality of life (EQ-5D-5L), residual symptoms, psychological distress (Hospital Anxiety and Depression Scale), and vocational outcomes (Work Ability Score) will be collected for all patients at the 12-month follow-up moment, as part of routine care, in accordance with Dutch and international stroke guidelines. 22-24 In case a patient reports headache, fatigue, or cognitive impairment, standardized questionnaires (Headache Impact Test-6, Fatigue Assessment Scale, and Checklist for Cognitive and Emotional Consequence of Stroke [CLCE-24; questions 1 to 13], respectively) will be collected to further evaluate the extent of these residual symptoms. The longterm VTE recurrence rate will be collected at 24 months after CVT diagnosis.

#### 5.3 Withdrawal of individual subjects

Subjects can leave the study at any time for any reason if they wish to do so without any consequences.

#### 5.4 Premature termination of the study

The study will be prematurely terminated if the Steering Committee decides this observational study is no longer clinically relevant, e.g. because new insights have rendered the research question irrelevant. In case of premature study termination, the results of the study thus far will be published as an exploratory report.

Version 3.1 - 13-08-2024 15 of 31

#### 6. STATISTICAL ANALYSES

Baseline characteristics will be presented for patients who are initially started on a DOAC and those who are initially started on VKA. Categorical data will be presented as counts and proportions, continuous data as means and standard deviations or medians and (interquartile) ranges, as appropriate. Missing data on confounders will be imputed using multiple imputation.

#### 6.1 Primary study endpoint

#### 6.1.1 Main analysis of primary endpoint

Comparisons will be made according to the intention-to-treat principle (i.e. according to the first oral anticoagulant that was started). Based on the results of the RESPECT CVT trial,<sup>9</sup> we expect an approximate 1.7% event rate for the primary outcome in the DOAC group and a 3.3% event rate in the VKA group, i.e. around 12 events in the total sample.

We will use propensity score inverse probability treatment weighting to calculate an adjusted odds ratio for the primary outcome. Based on the direct acyclic graph (Figure 3), the following confounders will be used to compute the propensity score:

- Age at time of CVT diagnosis
- ICH at CVT diagnosis, or after diagnosis but before start of oral anticoagulant treatment
- Glasgow Coma Scale at CVT diagnosis
- CNS infection concurrent with the index CVT
- Known antiphospholipid syndrome, or presence of antiphospholipid antibodies at start of oral anticoagulant treatment
- Cancer (defined as currently under treatment or diagnosed within 6 months prior to start of oral anticoagulant treatment)
- Previous VTE
- Previous major bleeding prior to the index CVT (according to ISTH criteria)
- Baseline renal function
- Concomitant antiplatelet use at start of oral anticoagulant treatment
- Country of inclusion's income group as classified by The World Bank.

Version 3.1 - 13-08-2024 16 of 31

We will analyze the balance of confounders among both treatment groups after propensity score inverse probability-weighting. A *last observation carried forward* approach will be used if the 6- or 12-month follow-up data are missing.



Figure 3. Directed Acyclic Graph depicting factors influencing anticoagulant treatment choice and risk of recurrent venous thrombotic event or major bleeding

#### 6.1.2 Sensitivity analyses for the primary endpoint

In addition to the main analysis of the primary endpoint, we will perform four sensitivity analyses for the primary endpoint. Firstly, we will perform a survival

Version 3.1 - 13-08-2024 17 of 31

analysis of the primary endpoint using the inverse probability weighting from the main analysis. Patients will be censored at the time of anticoagulant-switch or at the last follow-up moment (after 3, 6, or 12 months). Secondly, we will provide unadjusted analyses. Thirdly, we will repeat the analysis conducting a worst-case scenario approach i.e. using the assumption that all patients with missing outcome data would have suffered a primary endpoint event. Lastly, we will perform a descriptive ontreatment analysis.

#### 6.1.3 Subgroup analysis of primary endpoint

In an exploratory subgroup analysis, we will report all primary and secondary outcomes stratified by type of DOAC (i.e. apixaban, betrixaban, dabigatran, edoxaban, or rivaroxaban) if the number of cases is sufficient. In addition, we will perform a subgroup analysis for patients who were diagnosed with APS compared to patients who do not have APS. No formal statistical comparisons will be performed for these subgroup analyses.

#### 6.2 Secondary study parameter(s)

All secondary outcomes will be analysed with the same method as used for the main analysis. Confounders to be included in each propensity score calculation are detailed in Appendix C. Outcomes regarding the post-CVT residual symptoms and two-year VTE recurrence rate will be reported descriptively.

Version 3.1 - 13-08-2024 18 of 31

#### 7. ETHICAL CONSIDERATIONS

#### 7.1 Regulation statement

This study will be conducted in accordance with the principles of the Declaration of Helsinki, as amended by the World Medical Association General Assembly in October 2013, and with the guidelines for Good Clinical Practice.

#### 7.2 Recruitment and consent

The study uses only data that are collected as part of routine care. The local investigator at each participating center will inform eligible subjects of the study. All patients or their proxy's will be asked for written informed consent to allow use of their data in a coded manner in accordance with the European Union General Data Protection Regulation (GDPR) and other applicable laws for that particular hospital.

#### 7.3 Benefits and risks assessment

This study poses no risk and no burden to participants. Only existing patient care data will be used.

Version 3.1 - 13-08-2024 19 of 31

#### 8. ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION

#### 8.1 Handling, storage, and maintenance of data and documents

All patients will be assigned a unique study ID which contains no identifying information. Study data will be entered into the study database under this unique study ID by the local investigator. The study database will not contain directly identifying data such as name, address or date of birth. The subject identification code list linking the study ID with the source data remains at the local hospital and is stored by the local investigator separate from the study database. Only local investigators participating in the registry will have access to this list.

The study data will be kept for a minimum of 15 and a maximum of 25 years (conform the local requirements) after enrollment of the last patient into the registry.

The Amsterdam UMC will function as the controller of the data for this study. Castor Electronic Data Capture system will be used to collect all data in a standardized manner (www.castoredc.com). Amsterdam UMC has a data processor agreement with Castor EDC. Each center should comply with local laws and institutional rules regarding data storage and data transfer, sign the Data Transfer Agreement, and send the local IRB approval to the Study Coordinator before enrollment can start. Additional Data Transfer Agreements for the execution of substudies will be prepared as necessary.

#### 8.2 Study Oversight

The project leader has the final responsibility for the execution of the DOAC-CVT study. The Steering Committee will oversee the conduction of the study and provide support and guidance. The Steering Committee will meet twice a year, either in person or digitally. Additional Steering Committee meetings may be scheduled at the request of the Executive Committee. A national leader will be appointed by the Executive Committee for each country that participates in the study, and all national leaders are members of the Steering Committee. The Executive Committee supervises the day-to-day study execution for the Steering Committee. The day-to-day study execution will be coordinated by the study coordinator.

Version 3.1 - 13-08-2024 20 of 31

**Executive Committee** 

Dr. Jonathan Coutinho (project leader)

Amsterdam UMC, Amsterdam, the Netherlands

Dr. Jukka Putaala

Helsinki University Hospital, Helsinki, Finland

Prof. Jose Ferro

Hospital da Luz, University of Lisbon, Lisbon, Portugal

Prof. Turgut Tatlisumak

Sahlgrenska University Hospital, Gothenburg, Sweden

Dr. Diana Aguiar de Sousa

Centro Hospitalar Universitário Lisboa Central (ULS São José), Lisbon, Portugal

Dr. Katarina Jood

Sahlgrenska University Hospital, Gothenburg, Sweden

#### **Steering Committee**

Dr. Jonathan Coutinho

Amsterdam UMC, Amsterdam, the Netherlands

Dr. Jukka Putaala

Helsinki University Hospital, Helsinki, Finland

Prof. Jose Ferro

Hospital da Luz, University of Lisbon, Lisbon, Portugal

Prof. Turgut Tatlisumak

Sahlgrenska University Hospital, Gothenburg, Sweden

Drs. Mayte Sanchez van Kammen

Amsterdam UMC, Amsterdam, the Netherlands

Drs. Anita van de Munckhof

Amsterdam UMC, Amsterdam, the Netherlands

Dr. Diana Aguiar de Sousa

Centro Hospitalar Universitário Lisboa Central (ULS São José), Lisbon, Portugal

Dr. Katarina Jood

Sahlgrenska University Hospital, Gothenburg, Sweden

All national leaders (see Appendix D)

#### **Independent Adjudication Committee**

Prof. Saskia Middeldorp, chair

Radboud UMC, Nijmegen, the Netherlands

Prof. Lia Neto

Hospital de Santa Maria, Lisbon, Portugal

Prof. Marcel Arnold

Bern University Hospital, Bern, Switzerland

Version 3.1 - 13-08-2024 21 of 31

#### 8.3 Public disclosure and publication policy

This study is registered at clinicaltrials.gov and the study protocol has been published in a peer-reviewed journal.<sup>25</sup> A first draft of the main study paper will be drafted by the Executive Committee together with a PhD student. All Steering Committee members will be co-authors on the main study paper. All other investigators will be listed on the main study paper as members of the DOAC-CVT study group. In addition, participating centres may contribute one additional co-author after inclusion of 10 patients, and an additional co-author for each additional 20 patients included afterwards. All authors must fulfil the ICMJE criteria for scientific authorship. After publication of the primary study results, each participating investigator may submit proposals for a substudy to the Executive Committee. After approval by the Executive Committee, the local investigator of that hospital may take the lead in the execution and authorship of that particular substudy.

Version 3.1 - 13-08-2024 22 of 31

#### References

- 1. Silvis SM, de Sousa DA, Ferro JM, Coutinho JM. Cerebral venous thrombosis. *Nat Rev Neurol*. 2017;13(9):555-565. doi:10.1038/nrneurol.2017.104
- 2. Ferro JM, Canhao P, Stam J, Bousser MG, Barinagarrementeria F. Prognosis of cerebral vein and dural sinus thrombosis: results of the International Study on Cerebral Vein and Dural Sinus Thrombosis (ISCVT). *Stroke*. Mar 2004;35(3):664-70. doi:10.1161/01.Str.0000117571.76197.26
- 3. Coutinho JM, Zuurbier SM, Stam J. Declining mortality in cerebral venous thrombosis: a systematic review. *Stroke*. May 2014;45(5):1338-41. doi:10.1161/STROKEAHA.113.004666 4. Coutinho J, de Bruijn SF, Deveber G, Stam J. Anticoagulation for cerebral venous sinus thrombosis. *The Cochrane database of systematic reviews*. Aug 10 2011;(8):Cd002005. doi:10.1002/14651858.CD002005.pub2
- 5. Ferro JM, Bousser MG, Canhao P, et al. European Stroke Organization guideline for the diagnosis and treatment of cerebral venous thrombosis endorsed by the European Academy of Neurology. *Eur J Neurol*. Oct 2017;24(10):1203-1213. doi:10.1111/ene.13381 6. Saposnik G, Barinagarrementeria F, Brown RD, Jr., et al. Diagnosis and management of cerebral venous thrombosis: a statement for healthcare professionals from the American Heart Association/American Stroke Association. *Stroke*. Apr 2011;42(4):1158-92. doi:10.1161/STR.0b013e31820a8364
- 7. Foerch C, Lo EH, van Leyen K, Lauer A, Schaefer JH. Intracerebral Hemorrhage Formation Under Direct Oral Anticoagulants. *Stroke*. Apr 2019;50(4):1034-1042. doi:10.1161/STROKEAHA.118.023722
- 8. Vinogradova Y, Coupland C, Hill T, Hippisley-Cox J. Risks and benefits of direct oral anticoagulants versus warfarin in a real world setting: cohort study in primary care. *BMJ*. Jul 4 2018;362:k2505. doi:10.1136/bmj.k2505
- 9. Ferro JM, Coutinho JM, Dentali F, et al. Safety and Efficacy of Dabigatran Etexilate vs Dose-Adjusted Warfarin in Patients With Cerebral Venous Thrombosis: A Randomized Clinical Trial. *JAMA Neurol*. Sep 3 2019;doi:10.1001/jamaneurol.2019.2764
- 10. Lurkin A, Derex L, Fambrini A, Bertoletti L, Epinat M, Mismetti P, Dargaud Y. Direct Oral Anticoagulants for the Treatment of Cerebral Venous Thrombosis. *Cerebrovascular diseases (Basel, Switzerland)*. 2019;48(1-2):32-37. doi:10.1159/000502454
- 11. Rusin G, Wypasek E, Papuga-Szela E, Żuk J, Undas A. Direct oral anticoagulants in the treatment of cerebral venous sinus thrombosis: a single institution's experience. *Neurologia i neurochirurgia polska*. 2019;53(5):384-387. doi:10.5603/PJNNS.a2019.0037
- 12. Wasay M, Khan M, Rajput HM, et al. New Oral Anticoagulants versus Warfarin for Cerebral Venous Thrombosis: A Multi-Center, Observational Study. *J Stroke*. May 2019;21(2):220-223. doi:10.5853/jos.2019.00150
- 13. Lee GKH, Chen VH, Tan CH, et al. Comparing the efficacy and safety of direct oral anticoagulants with vitamin K antagonist in cerebral venous thrombosis. *J Thromb Thrombolysis*. Apr 11 2020;doi:10.1007/s11239-020-02106-7
- 14. Yaghi S, Shu L, Bakradze E, et al. Direct Oral Anticoagulants Versus Warfarin in the Treatment of Cerebral Venous Thrombosis (ACTION-CVT): A Multicenter International Study. *Stroke*. Mar 2022;53(3):728-738. doi:10.1161/STROKEAHA.121.037541 15. Field TS, Dizonno V, Almekhlafi MA, et al. Study of Rivaroxaban for
- Cerebral Venous Thrombosis: A Randomized Controlled Feasibility Trial Comparing Anticoagulation With Rivaroxaban to Standard-of-Care in Symptomatic Cerebral Venous Thrombosis. *Stroke*. Nov 2023;54(11):2724-2736. doi:10.1161/STROKEAHA.123.044113
- 16. Hiltunen S, Putaala J, Haapaniemi E, Tatlisumak T. Long-term outcome after cerebral venous thrombosis: analysis of functional and vocational outcome, residual symptoms, and adverse events in 161 patients. *J Neurol*. Mar 2016;263(3):477-84. doi:10.1007/s00415-015-7996-9
- 17. Koopman K, Uyttenboogaart M, Vroomen PC, van der Meer J, De Keyser J, Luijckx GJ. Long-term sequelae after cerebral venous thrombosis in functionally independent patients. *J Stroke Cerebrovasc Dis*. May-Jun 2009;18(3):198-202. doi:10.1016/j.jstrokecerebrovasdis.2008.10.004

- 18. Dentali F, Poli D, Scoditti U, et al. Long-term outcomes of patients with cerebral vein thrombosis: a multicenter study. Article. *J Thromb Haemost*. Jul 2012;10(7):1297-302. doi:10.1111/j.1538-7836.2012.04774.x
- 19. Schulman S, Kearon C. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. *J Thromb Haemost*. Apr 2005;3(4):692-4. doi:10.1111/j.1538-7836.2005.01204.x
- 20. Kaatz S, Ahmad D, Spyropoulos AC, Schulman S. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. *J Thromb Haemost*. Nov 2015;13(11):2119-26.
- 21. Aguiar de Sousa D, Lucas Neto L, Arauz A, et al. Early Recanalization in Patients With Cerebral Venous Thrombosis Treated With Anticoagulation. *Stroke*. Apr 2020;51(4):1174-1181. doi:10.1161/strokeaha.119.028532
- 22. Winstein CJ, Stein J, Arena R, et al. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. *Stroke*. Jun 2016;47(6):e98-e169. doi:10.1161/STR.0000000000000098
- 23. Lindsay MP, Norrving B, Furie KL, Donnan G, Langhorne P, Davis S. Global Stroke Guidelines and Action Plan: A Road Map for Quality Stroke Care. 2016. Accessed 5 March 2024. <a href="https://www.world-stroke.org/what-we-do/education-and-research/improving-access-to-quality-stroke-care/global-stroke-services-guideline-action-plan">https://www.world-stroke.org/what-we-do/education-and-research/improving-access-to-quality-stroke-care/global-stroke-services-guideline-action-plan</a>
- 24. Federatie Medisch Specialisten. Herseninfarct en hersenbloeding. Accessed 7 March 2024,
- https://richtlijnendatabase.nl/richtlijn/herseninfarct en hersenbloeding/startpagina herseninfarct -bloeding.html
- van de Munckhof A, Sanchez van Kammen M, Krzywicka K, et al. Direct oral anticoagulants for the treatment of cerebral venous thrombosis a protocol of an international phase IV study. *Front Neurol*. 2023;14:1251581. doi:10.3389/fneur.2023.1251581

Version 3.1 - 13-08-2024 24 of 31

#### APPENDIX A.

#### Standard Operating Procedure for the Scoring of Cerebral Venous Recanalization

[Standard Operating Procedure for Recanalization Assessment]

#### APPENDIX B.

#### ISTH definitions of major and clinically relevant non-major bleeding

#### Major bleeding<sup>19</sup>

Symptomatic presentation and

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells

#### Clinically relevant non-major bleeding<sup>20</sup>

Any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:

- Requiring medical intervention by a healthcare professional
- Leading to hospitalization or increased level of care
- Prompting a face to face (i.e., not just a telephone or electronic communication)
   evaluation

Version 3.1 - 13-08-2024 25 of 31

#### APPENDIX C.

All secondary outcomes at 6 months will be analysed with the same method as used in the main analysis. Confounders to be included in each propensity score calculation are listed below per outcome:



Figure 6. Directed Acyclic Graph depicting factors influencing anticoagulant treatment choice and risk of recurrent venous thrombotic event

Symptomatic recurrent VTE rate (Figure 6)

- Age at time of CVT diagnosis
- · GCS at CVT diagnosis
- Previous VTE

Version 3.1 - 13-08-2024 26 of 31



Figure 7. Directed Acyclic Graph depicting factors influencing anticoagulant treatment choice and risk of major or clinically relevant non-major bleeding

Major bleeding rate<sup>14</sup> (Figure 7)

- Age at CVT diagnosis
- CNS infection concurrent with the index CVT
- ICH at CVT diagnosis, or after diagnosis but before start of oral anticoagulant treatment
- Previous major bleeding prior to the index CVT (according to ISTH criteria)<sup>14</sup>

Clinically relevant non-major bleeding rate<sup>15</sup> (Figure 7)

- Age at CVT diagnosis
- CNS infection concurrent with the index CVT

Version 3.1 - 13-08-2024 27 of 31

- ICH at CVT diagnosis, or after diagnosis but before start of oral anticoagulant treatment
- Previous major bleeding prior to the index CVT (according to ISTH criteria)<sup>14</sup>



Figure 8. Directed Acyclic Graph depicting factors influencing anticoagulant treatment choice and risk of death or dependency<sup>2</sup>

#### All-cause mortality (Figure 8)

- Age at CVT diagnosis
- CNS infection concurrent with the index CVT
- · GCS at CVT diagnosis
- ICH at CVT diagnosis, or after diagnosis but before start of oral anticoagulant treatment

Version 3.1 - 13-08-2024 28 of 31

Modified Rankin Scale score (Figure 8)

- Age at CVT diagnosis
- CNS infection concurrent with the index CVT
- GCS at CVT diagnosis
- ICH at CVT diagnosis, or after diagnosis but before start of oral anticoagulant treatment



Figure 9. Directed Acyclic Graph depicting factors influencing anticoagulant treatment choice and risk of arterial thrombotic event

Arterial thrombotic events (Figure 9)

- Age at CVT diagnosis
- History of hypertension (as determined by treating physician)

Version 3.1 - 13-08-2024 29 of 31



Figure 10. Directed Acyclic Graph depicting factors influencing anticoagulant treatment choice and cerebral venous recanalization<sup>17</sup>

Cerebral venous recanalization rate (Figure 10)

- Age at CVT diagnosis
- Sex
- Isolated superior sagittal sinus thrombosis at diagnosis

Version 3.1 - 13-08-2024 30 of 31

APPENDIX D.

List of National Leaders of the DOAC-CVT study

| Country | National Leader | E-mail address |
|---|---|---|
| Argentina | Matías Alet | matias.alet@gmail.com |
| Australia | Timothy J. Kleinig | timothy.kleinig@sa.gov.au |
| Belgium | Robin Lemmens | robin.lemmens@uzleuven.be |
| Brazil | Adriana B. Conforto | adriana.conforto@gmail.com |
| Chile | Daniel Galdames Contreras | dgaldames@hcuch.cl |
| China | Xunming Ji | jixm@ccmu.edu.cn |
| Costa Rica | Miguel A. Barboza | miguel.barboza_e@ucr.ac.cr |
| Finland | Jukka Putaala | jukka.putaala@hus.fi |
| Germany | Sven Poli | sven.poli@uni-tuebingen.de |
| India | Sanjith Aaron | drsanjith@yahoo.co.uk |
| Israel | Ronen R. Leker | leker@hadassah.org.il |
| Italy | Francesco Dentali | fdentali@libero.it |
| Mexico | Antonio Arauz | antonio.arauz@prodigy.net.mx |
| the Netherlands | Jonathan M. Coutinho | j.coutinho@amsterdamumc.nl |
| New Zealand | Teddy Wu | teddyyhwu@gmail.com |
| Norway | Espen S. Kristoffersen | e.s.kristoffersen@medisin.uio.no |
| Pakistan | Mohammad Wasay | mohammad.wasay@aku.edu |
| Portugal | Diana Aguiar de Sousa | dianasousa@campus.ul.pt |
| Romania | Florina Antochi | flrant@yahoo.com |
| Spain | María Hernandez-Perez | mhernandez@igtp.cat |
| Sweden | Katarina Jood | katarina.jood@neuro.gu.se |
| Switzerland | Mirjam R. Heldner | mirjam.heldner@insel.ch |
| Turkey | Nilufer Yesilot | niluferyes@yahoo.com |
| United States | Wayneho Kam | wayneho.kam@duke.edu |

Version 3.1 - 13-08-2024 31 of 31